CLINICAL TRIAL: NCT06551376
Title: IVF CYCLE SCHEDULING WITH LATE LUTEAL PHASE VS. CONVENTIONAL EARLY FOLLICULAR PHASE START TO AVOID WEEKENDS RETRIEVALS: PROOF OF CONCEPT
Brief Title: LATE LUTEAL PHASE VS. CONVENTIONAL EARLY FOLLICULAR PHASE START IN IVF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinia de fertilización Asistida en el Hospital ABC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPI010924
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: IVF
Keywords: Ovarian Stimulation; luteal phase start; early follicular phase start; ovarian response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Follicular Phase ovarian stimulation (Placebo Comparator): Twenty patients started controlled ovarian stimulation (COS) after spontaneous menses
  Interventions: Other: Ovarian Stimulation Start
- Late Luteal Phase ovarian stimulation (Active Comparator): Twenty patients started stimulation on the Friday previous to a spontaneous menses (at the end of late luteal phase), regardless of cycle day.
  Interventions: Other: Ovarian Stimulation Start

INTERVENTIONS:
Other: Ovarian Stimulation Start — To compare ovarian response accordin to ovarian stimualtion start

SUMMARY:
To compare cycle outcomes after scheduling with the standard early follicular phase (EFP) versus late luteal phase (LLP) in patients undergoing GnRH antagonist cycles.

DETAILED DESCRIPTION:
Objective To compare cycle outcomes after scheduling with the standard early follicular phase (EFP) versus late luteal phase (LLP) in patients undergoing GnRH antagonist cycles.

Design Multicentric prospective non-randomized study

Setting Two university-affiliated private assisted reproduction centers.

Patient(s) Regularly cycling women aged ≤40 years with fewer than one previous IVF attempts were enrolled. Previous low responses to controlled ovarian hyperstimulation, ovarian surgery, or polycystic ovary were exclusion criteria.

Intervention(s) Twenty patients started controlled ovarian stimulation (COS) after spontaneous menses; similarly, twenty patients started stimulation on the Friday previous to a spontaneous menses (at the end of late luteal phase), regardless of cycle day.

Main Outcome Measure(s) Primary outcome: number of mature oocytes retrieved. Secondary outcomes: fertilization rate, viable embryo rate per oocyte retrieved, cancellation rate, and clinical pregnancy outcomes from FET cycles.

ELIGIBILITY:
Inclusion Criteria:

* Regularly cycling women aged ≤40 years with fewer than one previous IVF attempts were enrolled

Exclusion Criteria:

* Previous low responses to controlled ovarian hyperstimulation, ovarian surgery, or polycystic ovary were exclusion criteria

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
mature oocytes retrieved | At retrieval

SECONDARY OUTCOMES:
fertilization rate | 24 hours after retrieval
viable embryo rate per oocyte retrieved | 5 days after retrieval
cancellation rate | 14 days after cycle start

IPD SHARING:
Plan to Share IPD: Undecided